CLINICAL TRIAL: NCT03202550
Title: Oral Sedation During Cervical Dilator Placement: A Randomized Controlled Trial
Brief Title: Oral Sedation During Cervical Dilator Placement
Acronym: OSDI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00117627
Record Dates: First submitted 2017-06-27; First posted 2017-06-28 (Actual); Results first posted 2020-03-06 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Oral Sedation and Cervical Dilator Pain
Keywords: Oral Sedation; Lorazepam; Oxycodone
MeSH Terms: interventions — Oxycodone; Lorazepam

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participant, provider, and nursing staff will be blinded to the intervention. The pharmacy will prepare the treatment drugs and placebos.. Randomization will be stratified by gestational age (>= 20 weeks or <20 weeks) and the randomization allocation sequence will be computer-generated with a random number generator by a statistician. The pharmacist will be aware of the randomization sequence and will dispense the drugs as appropriate, while keeping track of which arms participants were randomized to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo Arm (Placebo Comparator): Two oral placebo pills (microcrystalline cellulose capsules)
  Interventions: Drug: Placebo Comparator
- Active Drug Arm: Lorazepam and Oxycodone (Active Comparator): 1 mg of oral lorazepam and 5 mg of oral oxycodone (also encased in microcrystalline cellulose capsules)
  Interventions: Drug: Oxycodone and Lorazepam (Active Comparator)

INTERVENTIONS:
Drug: Oxycodone and Lorazepam (Active Comparator) — Oxycodone and Lorazepam
  Other Names: Oral Oxycodone; Oral Lorazepam; Ativan; OxyIR; Roxicodone
  Arms: Active Drug Arm: Lorazepam and Oxycodone
Drug: Placebo Comparator — Placebo oral pills
  Arms: Placebo Arm

SUMMARY:
This will be a randomized, double-blind, placebo-controlled trial involving 2 arms. It will be comparing the effects of placebo compared to 1 mg oral lorazepam/5 mg oral oxycodone on pain scores during cervical dilator placement prior to dilation and evacuation (D&E).

DETAILED DESCRIPTION:
Potential participants will be first introduced to the study via routine intake call. Participants will be identified at the participant's office visits to the Johns Hopkins' Women's Center for Family Planning. If a patient desires D&E for a second trimester pregnancy, the patient will first receive standard counseling. Only after providing written informed consent for the procedure will the patients be screened for eligibility in the study. If the patient is eligible the participant will be asked by a member of the research team if the patient is interested in participating. If the patient is, the study will be explained to the participant and written consent will be obtained after participant is given the opportunity to have all questions answered.

The study is randomized, double-blind, placebo-controlled trial involving 2 arms. Participants will first complete a survey to collect demographic data.

Participants in both arms will receive the institution's current standard analgesia for cervical dilator placement. In addition to this standard regimen, participants will be randomized to receive either: (1) a dose of two oral placebo pills, or (2) 1mg of oral lorazepam with 5 mg of oral oxycodone prior to cervical dilator placement.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-50 years
* English speaking
* With an intrauterine pregnancy (either viable or non-viable) between the gestational ages of 17w0d and 23w6d
* Have a support person present with participant
* Have a cell phone capable of text messaging (optional)

Exclusion Criteria:

* Non-English-speaking
* Taking a daily benzodiazepine or opiate
* Have a known allergy or contraindication to NSAIDs, opiates, or benzodiazepines

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Sufrin, Principal Investigator — Johns Hopkins University; Jessica K Lee, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins' Women's Center for Family Planning, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The study plans to share placebo data (without PHI) with colleagues at University of California Davis at the end of the study. A Memorandum of Understanding will be created prior to sharing (MOU) and data will be shared across a secure server.

REFERENCES:
- [Background] Mercier RJ, Liberty A. Intrauterine lidocaine for pain control during laminaria insertion: a randomized controlled trial. Contraception. 2014 Dec;90(6):594-600. doi: 10.1016/j.contraception.2014.07.008. Epub 2014 Jul 23. PMID 25139724
- [Background] Soon, R. T., M.; Salcedo. J.; Kaneshiro, B., Paracervical block to decrease pain with second-trimester laminaria insertion: a randomized controlled trial. Contraception 2016, 94 (4), 389.
- [Background] Wong CY, Ng EH, Ngai SW, Ho PC. A randomized, double blind, placebo-controlled study to investigate the use of conscious sedation in conjunction with paracervical block for reducing pain in termination of first trimester pregnancy by suction evacuation. Hum Reprod. 2002 May;17(5):1222-5. doi: 10.1093/humrep/17.5.1222. PMID 11980742
- [Background] Wiebe E, Podhradsky L, Dijak V. The effect of lorazepam on pain and anxiety in abortion. Contraception. 2003 Mar;67(3):219-21. doi: 10.1016/s0010-7824(02)00516-4. PMID 12618257

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three participants who were enrolled but did not receive the intervention had either chosen not to proceed further with the study or were not able to swallow the study drugs.
Period: Overall Study
Arm/Group | Placebo Arm | Active Drug Arm: Lorazepam and Oxycodone
Started | 13 | 11
Completed | 13 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Arm | Active Drug Arm: Lorazepam and Oxycodone | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 11 | 24
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 12 | 11 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 10 | 21
  White | 1 | 0 | 1
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: Cervical Dilator Placement Pain as Assessed by VAS on a Tablet Device
Description: Compare pain scores on a 100 mm visual analog scale (VAS) (anchors 0=no pain; 100=worst pain ever)
Time Frame: Immediately after the last dilator is placed, up to 1 minute
Population: One participant in the active drug arm was determined to not need to have cervical dilators placed, so this participant was not included in the total number of active drug arm participants.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo Arm | Active Drug Arm: Lorazepam and Oxycodone
Number analyzed (Participants) | 13 | 10
units on a scale | 55 [33 to 82] | 44 [10 to 80]

2. Secondary Outcome: Number of Participants With Desired Number of Dilators Inserted
Description: Assess whether desired number of dilators was not able to be successfully inserted, comparing 2 arms.
Time Frame: After speculum removed, up to 30 minutes
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Arm | Active Drug Arm: Lorazepam and Oxycodone
Number analyzed (Participants) | 13 | 10
Participants | 13 | 10

3. Secondary Outcome: Baseline Pain Score Before Drugs Were Administered
Description: Compare pain scores on a 100 mm visual analog scale (VAS) (anchors 0=no pain; 100=worst pain ever)
Time Frame: pain score given prior to administration of study drugs, up to 1 minute
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo Arm | Active Drug Arm: Lorazepam and Oxycodone
Number analyzed (Participants) | 13 | 10
units on a scale | 3 [0 to 6] | 2 [0 to 12]

4. Secondary Outcome: Pain Score Before Speculum Placement
Description: Compare pain scores on a 100 mm visual analog scale (VAS) (anchors 0=no pain; 100=worst pain ever)
Time Frame: pain score given before specula placed, up to 1 minute
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo Arm | Active Drug Arm: Lorazepam and Oxycodone
Number analyzed (Participants) | 13 | 10
units on a scale | 1 [0 to 1] | 1 [0 to 2]

5. Secondary Outcome: Pain Score After Speculum Placement
Description: Compare pain scores on a 100 mm visual analog scale (VAS) (anchors 0=no pain; 100=worst pain ever)
Time Frame: pain score given at time of speculum placement, up to 1 minute
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo Arm | Active Drug Arm: Lorazepam and Oxycodone
Number analyzed (Participants) | 13 | 10
units on a scale | 20 [12 to 43] | 11 [3 to 51]

6. Secondary Outcome: Pain Score at Tenaculum Placement
Description: Compare pain scores on a 100 mm visual analog scale (VAS) (anchors 0=no pain; 100=worst pain ever)
Time Frame: Immediately scored at time of tenacula placement, up to 1 minute
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo Arm | Active Drug Arm: Lorazepam and Oxycodone
Number analyzed (Participants) | 13 | 10
units on a scale | 31 [15 to 56] | 50 [2 to 70]

7. Secondary Outcome: Pain Score During Paracervical Block
Description: Compare pain scores on a 100 mm visual analog scale (VAS) (anchors 0=no pain; 100=worst pain ever)
Time Frame: pain score given at time of paracervical block administration, up to 1 minute
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo Arm | Active Drug Arm: Lorazepam and Oxycodone
Number analyzed (Participants) | 13 | 10
units on a scale | 57 [16 to 69] | 51 [6 to 71]

8. Secondary Outcome: Pain Score After First Dilator Placement
Description: Compare pain scores on a 100 mm visual analog scale (VAS) (anchors 0=no pain; 100=worst pain ever)
Time Frame: pain score given immediately after first dilator placed, up to 1 minute
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo Arm | Active Drug Arm: Lorazepam and Oxycodone
Number analyzed (Participants) | 13 | 10
units on a scale | 50 [16 to 56] | 9 [2 to 52]

9. Secondary Outcome: Pain Score 15 Minutes After Last Dilator Placed
Description: Compare pain scores on a 100 mm visual analog scale (VAS) (anchors 0=no pain; 100=worst pain ever). This was to be assessed at 15 minutes after last dilator is placed. Some participants had this assessment done up to 45 minutes after last dilator was placed because it could not be done at 15 minutes (some were being attended to by a nurse at the 15 minutes mark).
Time Frame: Assessed up to 45 minutes after last dilator placed
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo Arm | Active Drug Arm: Lorazepam and Oxycodone
Number analyzed (Participants) | 13 | 10
units on a scale | 29 [14 to 44] | 13 [0 to 49]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from subjects for the 1 day that they were enrolled and active in the study.
Arm/Group | Placebo Arm | Active Drug Arm: Lorazepam and Oxycodone
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 1/13 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Arm (N=13) | Active Drug Arm: Lorazepam and Oxycodone (N=11)
Cervical laceration (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Laceration occurred when tenaculum was placed on cervix

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-17): https://cdn.clinicaltrials.gov/large-docs/50/NCT03202550/Prot_SAP_000.pdf